CLINICAL TRIAL: NCT07394920
Title: The Role of Sodium Bicarbonate Enema in Improving Constipation and Reducing Uremic Toxins in Chronic Kidney Disease Patients.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Goubara Abdulhaq, residant doctor at Assiut university hospital, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sodium bicarbonate enema CKD
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Active Comparator): patients with CKD will recived sodium bicarbonate enema
  Interventions: Procedure: sodium bicarbonate enema

INTERVENTIONS:
Procedure: sodium bicarbonate enema — patients with CKD will recived sodium bicarbonate enema

SUMMARY:
Chronic kidney disease (CKD) is a progressive condition characterized by a gradual loss of kidney function, often resulting in the accumulation of metabolic waste products. One of the emerging areas of interest in CKD management is the gut-kidney axis, which highlights the interplay between gut microbiota and renal health. CKD patients frequently exhibit gut dysbiosis and increased production of gut-derived uremic toxins such as indoxyl sulfate and p-cresyl sulfate, which can further exacerbate kidney damage and systemic inflammation.

CKD causes acidosis because damaged kidneys can't effectively excrete acids from the body or produce enough bicarbonate to neutralize them. This imbalance leads to a buildup of acids in the blood, resulting in metabolic acidosis, where acid levels in the blood become greater than normal.

Recent evidence suggests a close association between constipation and clinical outcomes such as cardiovascular disease, CKD progression and mortality(1-4). In particular, numerous observational studies have reported a higher prevalence of constipation in patients with CKD. Although the global prevalence of constipation in the general population has been estimated at approximately 14%, the prevalence in patients with CKD is reported to be much higher(5). A recent meta analysis reported a constipation prevalence of 38.8% in patients with advanced non-dialysis CKD(6). Patients with end-stage renal disease (ESRD) have been shown to have a substantially higher constipation prevalence, with some studies reporting over 50%(7).

This study focuses on using the GIT as an additional excretory pathway of the uremic toxins via using sodium bicarbonate enema in patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

* - Adults aged 18-60 years
* Diagnosed with CKD stage 3-4
* Stable renal function for 3 months
* Able to give informed consent

Exclusion Criteria:

* - Active GI disease (IBD, colon cancer, severe hemorrhoids, anal fissure)
* Recent abdominal or colorectal surgery
* Severe cardiovascular conditions
* Pregnancy or breastfeeding
* Electrolyte imbalance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
uremic toxins level | 3 months
  uremic toxins level after sodium bicarbonate enema